CLINICAL TRIAL: NCT06645379
Title: Application of Platelet-rich Plasma (PRP) in Reproductive Medicine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-176
Record Dates: First submitted 2024-10-07; First posted 2024-10-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Premature Ovarian Insufficiency; Intrauterine Adhesion; Poor Ovarian Response; Repeated Implantation Failure; Thin Endometrium
MeSH Terms: conditions — Primary Ovarian Insufficiency; Gynatresia | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- reproductive disease (Experimental): Platelet-rich Plasma injection
  Interventions: Other: Platelet-Rich Plasma (PRP) Injections

INTERVENTIONS:
Other: Platelet-Rich Plasma (PRP) Injections — Transvaginal or laparoscopic injection for ovarian diseases (Premature ovarian insufficiency and Poor ovarian response). Intrauterine perfusion or sub-endometrium injection for uterine diseases (intrauterine adhesion, thin endometrium, and repeated implantation failure)

SUMMARY:
Female fertility is affected by many factors, such as ovarian function, fallopian tube patency, uterine environment, and mental state, among which the ovaries and endometrium are more important. In reproductive medicine, ovarian dysfunction, poor ovarian reaction, intrauterine adhesion, recurrent implantation failure, and thin endometrium are the five most common diseases that affect fertility. These five diseases lack effective treatment, and previous studies have shown that platelet-rich plasma is promising in treating these five diseases, so it is necessary to further explore the therapeutic effect and potential mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Premature ovarian insufficiency: ① Women aged >18 and <40 years old; ② Oligomenorrhea or amenorrhea for more than 4 months (excluding pregnancy); ③ Basal follicle stimulating hormone (FSH) >25IU/L (interval >4 weeks) at least 2 times, or total antral follicles (AFC) <5, or anti-Mullerian hormone (AMH) <1.1ng/mL.
* Poor ovarian response: ① Advanced age (≥40 years) or other risk factors for poor ovarian response; ② Poor ovarian response in previous IVF cycle, with ≤3 oocytes retrieved using conventional protocols; ③ Decreased ovarian reserve (antral follicle count <5~7 or anti-Müllerian hormone <0.5~1.1 ug/L). Meeting any 2 of the above 3 criteria is sufficient.
* Intrauterine adhesion: ① Diagnosed by hysteroscopy and scored ≥5 points according to the American Fertility Society criteria (1988); ② With symptoms such as reduced menstrual flow amenorrhea, periodic lower abdominal pain, infertility, or recurrent miscarriage; ③ Adult women with the desire to conceive.
* Thin endometium: ①Endometrial thickness <7mm on ovulation day or on the day of human chorionic gonadotropin (HCG) injection, or <7mm on progesterone conversion day when using conventional hormone replacement therapy, ②adult women with the desire to comceive.
* Repeated implantation failure: Women under 40 years old who have failed to achieve clinical pregnancy after transplanting at least three high-quality embryos within three fresh or frozen cycles. High-quality embryos include: Day 3 embryos (with ≥8 cells, evenly sized blastomeres, and <10% fragmentation) and blastocysts (≥3BB).

Exclusion Criteria:

* Alanine aminotransferase > 3 times the normal upper limit or estimated glomerular filtration rate (EGFR) < 90 ml/min;
* Suffering from hemorrhagic diseases (such as hemophilia) or taking anticoagulant or antiplatelet drugs;
* Suffering from serious mental illness, cardiovascular and cerebrovascular diseases and malignant tumors;
* Suffering from diabetes with poor blood sugar control or other systemic diseases;
* Drug abuse, alcoholism or drug addiction;
* Participated in other interventional clinical studies within half a year;
* Poor compliance;
* Other circumstances that are not suitable for participating in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
adverse events or serious adverse events | From enrollment to the end of treatment at 3 months
  Discomfort or clinically significant abnormalities reported by patients after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided